CLINICAL TRIAL: NCT05310526
Title: Implementation of the Brazilian Cardioprotective Diet in Primary Health Care: a Cluster Randomized Type II Hybrid Implementation Study
Brief Title: BALANCE Diet Implementation in Primary Health Care: a Cluster Randomized Type II Hybrid Implementation Study
Acronym: Implementa-MAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Implementa-MAC
Record Dates: First submitted 2022-03-16; First posted 2022-04-05 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Obesity; Hypertension; Diabetes; Dyslipidemias
MeSH Terms: conditions — Obesity; Hypertension; Diabetes Mellitus; Dyslipidemias | interventions — Sensitivity Training Groups

STUDY DESIGN:
Intervention Model Description: Cluster-Randomized Trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): 1. Distribution of the Brazilian cardioprotective diet manual to primary health care
  2. Training to prescribe the cardioprotective Brazilian diet. the training consists of 5 face-to-face modules lasting 4 hours each, in addition to a virtual module and group exercises.
  3. Audit feedback
  Interventions: Other: Training Group
- Control Group (No Intervention): Distribution of the Brazilian cardioprotective diet manual to primary health care professionals

INTERVENTIONS:
Other: Training Group — Training for prescribing the Brazilian cardioprotective diet
  Arms: Intervention Group

SUMMARY:
This is an implementation type II hybrid study with randomisation in cluster, whose objective is to compare two strategies of implementation of the Brazilian cardioprotective diet guidelines in primary health care in two Brazilian cities. All health professionals from the health units (clusters) randomized to the intervention group will receive training on the subject. The health professionals from the health units randomized to the control group will follow the usual activities, receiving only the printed guidelines, as usually done. After 6 months, the prescription rate of the Brazilian cardioprotective diet will be evaluated, as well as the quality of the diet of patients in both groups.

ELIGIBILITY:
Clusters Inclusion criteria: All Public Primary Care Units from both cities will be included. However, the Health services that encourage health professionals to use the Cardioprotective Food manual before randomization will be excluded.

Participants (patients) Inclusion criteria:

* Individuals aged ≥20 years of either sex who have a previous medical diagnosis of at least one of the following conditions:
* Type 2 diabetes mellitus;
* Systemic arterial hypertension (Systolic blood pressure ≥140 mmHg or diastolic blood pressure greater than ≥90 mmHg or in drug treatment for hypertension);
* Isolated hypercholesterolemia: isolated increase in LDL-c (LDL-c ≥ 160 mg/dL).
* Isolated hypertriglyceridemia: isolated increase in triglycerides (TG ≥ 150 mg/dL or ≥ 175 mg/dL if the sample is obtained without fasting).
* Obesity or overweight (body mass index ≥25.0 kg/m2).

Exclusion Criteria:

* Prior cardiovascular event (acute myocardial infarction, stroke, peripheral arterial disease);
* Psychiatric or neurocognitive condition that prevents understanding of guidelines (defined by the clinical judgment of the investigators);
* Life expectancy less than 6 months (example: metastatic malignant neoplasm) to be defined by the investigator's judgment;
* Pregnancy or lactation;
* Liver failure with a previous history of encephalopathy or anasarca;
* Chronic renal failure;
* Organ transplantation;
* Gastroplasty for less than a year;
* Impossibility of oral feeding.
* No access to internet or mobile phone.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 786 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
Brazilian cardioprotective diet prescription rate | 6 months
  Implementation Primary Outcome (rate of eligible individuals who received Brazilian cardioprotective diet prescription)
food intake of 400g of vegetables per day | 6 months
  Eficacy Primary Outcome - number of patients that achieve the goal of eating 400g of vegetable/day

SECONDARY OUTCOMES:
Implementing the extra dietaty guidelines | 6 months
  rate of eligible individuals who received extra dietaty guidelines
Professionals' understanding of the Brazilian cardioprotective diet | right after intervention and 6 months after intervenions.
  standardized questionnaire. Continuous result (number of correct answers) and dichotomous (good knowledge / poor knowledge)
Patients' understanding of the Brazilian cardioprotective diet | right after intervention and 6 months after intervenions.
  standardized questionnaire. Continuous result (number of correct answers) and dichotomous (good knowledge / poor knowledge)
Patients' adherence to dietary guidelines | right after intervention and 6 months after intervenions.
  Vigitel dietary indicators
Participants' weight | right after intervention and 6 months after intervenions.
  wheight in kg
Barriers and facilitators identified in the implementation of the Brasilian Cardioprotective diet in health facilities (situational diagnosis). | 6 months
  Qualitative metodology: Focus groups with stakeholdrs and professionals involved in the implementation processo to identify barriers and facilitators perceived by them
Professionals' perception regarding the incorporation of MAC guidelines into practice (implementation component) | right after intervention and 6 months after intervenions.
  standardized questionnaire. Dichotomus result (Agree/Disagree with the incorporation)

CONTACTS AND LOCATIONS:
Locations (1):
- Prefeitura Municipal de Foz do Iguaçu, Foz do Iguaçu, Brazil

IPD SHARING:
Plan to Share IPD: Undecided